CLINICAL TRIAL: NCT00002171
Title: A Phase II, Randomized, Placebo-Controlled Study of the Safety and Efficacy of Viracept in Combination With Antiretroviral Therapy in HIV Positive Women With <= 1 Month of Prior Treatment With d4T and/or 3TC
Brief Title: A Study of Viracept in HIV-Positive Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agouron Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 259D; Study 534; AG1343 - 534
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-05

CONDITIONS: HIV Infections
Keywords: Placebos; Drug Therapy, Combination; Stavudine; HIV Protease Inhibitors; Lamivudine; Nelfinavir; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir mesylate

SUMMARY:
The purpose of this study is to see if it is safe and effective to give Viracept plus stavudine (d4T) plus lamivudine (3TC) to HIV-positive women with a CD4 count <= 400 cells/mm3. This study also examines how the body handles Viracept when given with d4T and 3TC.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* CD4 T cell count <= 400 cells/mm3.

Exclusion Criteria

Prior Medication:

Excluded:

* Prior therapy or less than 1 month of therapy with d4T and/or 3TC.
* Prior protease inhibitor therapy.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Cntr, Los Angeles, California
  - HIV Outpatient Clinics / LA State Univ Med Ctr, New Orleans, Louisiana
  - Baylor Univ, Houston, Texas